CLINICAL TRIAL: NCT00743730
Title: Outcomes And Parent Satisfaction Associated With Parent/Nurse Controlled Analgesia In Pediatric Patients With Developmental Delay
Brief Title: Parent Nurse Controlled Analgesic in Pediatric Patients With Developmental Delay
Acronym: PNCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Michelle Czarnecki, Advanced Practice Nurse, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHW 05/02, HRRC 008-05
Record Dates: First submitted 2008-06-12; First posted 2008-08-29 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Post Operative Pain
Keywords: developmental delay; cognitive impairment; pain control; post operative pain; opioid; pain assessment; Parent Nurse controlled Analgesic; patient controlled analgesic; children; pain; analgesic; safety; parent satisfaction; nurse satisfaction; Pediatric
MeSH Terms: conditions — Pain, Postoperative; Learning Disabilities; Cognitive Dysfunction; Agnosia; Pain | interventions — Morphine; Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Active Comparator): Parent and Nurse Controlled Analgesics with basal
  Interventions: Other: Pain and standard side effect management for PNCA with basal method.
- II (Active Comparator): Parent and Nurse Controlled Analgesics without basal
  Interventions: Other: Pain and standard side effect management with PNCA without basal
- III (Active Comparator): Intermittent opioid administered IV on an "as needed" basis
  Interventions: Other: Pain and standard side effect management with IV on an as needed basis method.

INTERVENTIONS:
Other: Pain and standard side effect management for PNCA with basal method. — Comparing pain management and parent and nurse satisfaction with medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
  Other Names: PNCA with basal
  Arms: I
Other: Pain and standard side effect management with PNCA without basal — Comparing pain management and parent nurse satisfaction with pain mediation delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
  Other Names: PNCA without basal
  Arms: II
Other: Pain and standard side effect management with IV on an as needed basis method. — Comparing pain management and parent and nurse satisfaction with pain medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol.
  Other Names: morphine injection; pain medication administered by IV as needed
  Arms: III

SUMMARY:
The purpose of this study is to compare, the safety, efficacy and level of parent and nurse satisfaction with three methods of opioid administration post-operatively in children (4-18 years of age) with developmental delay.

DETAILED DESCRIPTION:
Children with developmental delay are at higher risk for inadequate pain assessment and management. Patient controlled analgesia (PCA) allows patients to administer opioids by pushing a PCA button when needed. This eliminates the delay of waiting for a nurse to obtain and administer pain medication. PCA has been shown to be safe, effective, and superior to intramuscular, intermittent opioid dosing for pain management in children. Often, children with developmental delays cannot operate a PCA independently, can not self report their pain and are often given pain medication "as needed" through an IV. Parent/Nurse Controlled Analgesia (PNCA) allows parents and nurses to push the PCA button for patients who are not able to do so themselves. This way of giving pain medicine has not been thoroughly studied. Some healthcare professionals use PNCA for these children, others do not. This study is being done to compare PNCA & intermittent opioid administration. Participants will be randomized into one of the three study groups:

1. Parent/Nurse controlled Analgesia (PNCA) with a continuous intravenous (IV)infusion of pain medicine.
2. PNCA without continuous IV infusion of pain medicine.
3. Pain medicine given through IV administered on an "as needed" basis(PRN) by the nurse.

The Acute Pain Service will follow all three groups of patients throughout the study. This team specializes in the management of children's pain. Pain team is also available 24 hours a day, 7 days a week. The study will continue until child can tolerate pain medication in his/her stomach.

Data will be collected regarding safety, efficacy, parent & Nurse satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Children with developmental delay between 4 and 18 years of age who are unable to operate PCA due to developmental delay.
* Children scheduled for surgery anticipated to require >24hour stay with anticipation of IV narcotics will be required.
* Children whose parents are able to verbalize an understanding of PNCA.
* Parents with fluency in english(both speaking and writing).

Exclusion Criteria:

* Patients who do not meet inclusion criteria
* Patients whose parents do not give informed consent
* patients allergic to both morphine and hydromorphone
* patients with severe physiologically altering obstructive sleep apnea
* Patients who are or are expected to remain on a ventilator
* Patients receiving an epidural -

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2005-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Czarnecki, MSN RN CPNP, Principal Investigator — Childrens Hospital of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Doyle E, Harper I, Morton NS. Patient-controlled analgesia with low dose background infusions after lower abdominal surgery in children. Br J Anaesth. 1993 Dec;71(6):818-22. doi: 10.1093/bja/71.6.818. PMID 8280546
- [Background] Doyle E, Robinson D, Morton NS. Comparison of patient-controlled analgesia with and without a background infusion after lower abdominal surgery in children. Br J Anaesth. 1993 Nov;71(5):670-3. doi: 10.1093/bja/71.5.670. PMID 8251277
- [Background] Foster RL, Varni JW. Measuring the quality of children's postoperative pain management: initial validation of the child/parent Total Quality Pain Management (TQPM) instruments. J Pain Symptom Manage. 2002 Mar;23(3):201-10. doi: 10.1016/s0885-3924(01)00411-0. PMID 11888718
- [Background] Gaukroger PB, Tomkins DP, van der Walt JH. Patient-controlled analgesia in children. Anaesth Intensive Care. 1989 Aug;17(3):264-8. doi: 10.1177/0310057X8901700304. PMID 2774144
- [Background] Gureno MA, Reisinger CL. Patient controlled analgesia for the young pediatric patient. Pediatr Nurs. 1991 May-Jun;17(3):251-4. PMID 2062584
- [Background] Kotzer AM, Foster R. Children's use of PCA following spinal fusion. Orthop Nurs. 2000 Sep-Oct;19(5):19-27; quiz 28-30. doi: 10.1097/00006416-200019050-00005. PMID 11153382
- [Background] Malviya S, Voepel-Lewis T, Tait AR, Merkel S, Lauer A, Munro H, Farley F. Pain management in children with and without cognitive impairment following spine fusion surgery. Paediatr Anaesth. 2001 Jul;11(4):453-8. doi: 10.1046/j.1460-9592.2001.00686.x. PMID 11442864
- [Background] McGrath PJ, Rosmus C, Canfield C, Campbell MA, Hennigar A. Behaviours caregivers use to determine pain in non-verbal, cognitively impaired individuals. Dev Med Child Neurol. 1998 May;40(5):340-3. PMID 9630262
- [Background] McNeely JK, Trentadue NC. Comparison of patient-controlled analgesia with and without nighttime morphine infusion following lower extremity surgery in children. J Pain Symptom Manage. 1997 May;13(5):268-73. doi: 10.1016/s0885-3924(96)00324-7. PMID 9185432
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Miaskowski C, Crews J, Ready LB, Paul SM, Ginsberg B. Anesthesia-based pain services improve the quality of postoperative pain management. Pain. 1999 Mar;80(1-2):23-9. doi: 10.1016/s0304-3959(98)00192-4. PMID 10204714
- [Background] Oberlander TF, Gilbert CA, Chambers CT, O'Donnell ME, Craig KD. Biobehavioral responses to acute pain in adolescents with a significant neurologic impairment. Clin J Pain. 1999 Sep;15(3):201-9. doi: 10.1097/00002508-199909000-00007. PMID 10524473
- [Background] Pellino TA, Ward SE. Perceived control mediates the relationship between pain severity and patient satisfaction. J Pain Symptom Manage. 1998 Feb;15(2):110-6. PMID 9494309
- [Background] Peters JW, Bandell Hoekstra IE, Huijer Abu-Saad H, Bouwmeester J, Meursing AE, Tibboel D. Patient controlled analgesia in children and adolescents: a randomized controlled trial. Paediatr Anaesth. 1999;9(3):235-41. doi: 10.1046/j.1460-9592.1999.00358.x. PMID 10320603
- [Background] Rodgers BM, Webb CJ, Stergios D, Newman BM. Patient-controlled analgesia in pediatric surgery. J Pediatr Surg. 1988 Mar;23(3):259-62. doi: 10.1016/s0022-3468(88)80735-8. PMID 3357143
- [Background] Rusy, L. M., Olsen, D. J., & Farber, N. E. (1997). Successful use of patient-controlled analgesia in pediatric patients 2 and 3 years old: Two case reports. Am J Anesthesiol, 14(4), 212-214.
- [Background] Voepel-Lewis T, Merkel S, Tait AR, Trzcinka A, Malviya S. The reliability and validity of the Face, Legs, Activity, Cry, Consolability observational tool as a measure of pain in children with cognitive impairment. Anesth Analg. 2002 Nov;95(5):1224-9, table of contents. doi: 10.1097/00000539-200211000-00020. PMID 12401598
- [Background] Yildiz K, Tercan E, Dogru K, Ozkan U, Boyaci A. Comparison of patient-controlled analgesia with and without a background infusion after appendicectomy in children. Paediatr Anaesth. 2003 Jun;13(5):427-31. doi: 10.1046/j.1460-9592.2003.01061.x. PMID 12791117
- [Derived] Czarnecki ML, Hainsworth K, Simpson PM, Arca MJ, Uhing MR, Zhang L, Grippe A, Varadarajan J, Rusy LM, Firary M, Weisman SJ. A Pilot Randomized Controlled Trial of Outcomes Associated with Parent-Nurse Controlled Analgesia vs. Continuous Opioid Infusion in the Neonatal Intensive Care Unit. Pain Manag Nurs. 2020 Feb;21(1):72-80. doi: 10.1016/j.pmn.2019.08.002. Epub 2019 Sep 4. PMID 31494028
- [Derived] Czarnecki ML, Hainsworth KR, Simpson PM, Weisman SJ. Parent/Nurse-Controlled Analgesia Compared with Intravenous PRN Opioids for Postsurgical Pain Management in Children with Developmental Delay: A Randomized Controlled Trial. Pain Med. 2018 Apr 1;19(4):742-752. doi: 10.1093/pm/pnx257. PMID 29099960

RESULTS

PARTICIPANT FLOW:
Groups:
- PNCA With Basal: Parent and Nurse Controlled Analgesics with basal
  Pain and standard side effect management for PNCA with basal method.: Comparing pain management and parent and nurse satisfaction with medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
- PNCA w/o Basal: Parent and Nurse Controlled Analgesics without basal
  Pain and standard side effect management with PNCA without basal: Comparing pain management and parent nurse satisfaction with pain mediation delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
- Medication as Needed: Intermittent opioid administered IV on an "as needed" basis
  Pain and standard side effect management with IV on an as needed basis method.: Comparing pain management and parent and nurse satisfaction with pain medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol.
Period: Overall Study
Arm/Group | PNCA With Basal | PNCA w/o Basal | Medication as Needed
Started | 27 | 34 | 33
Completed | 22 | 30 | 28
Not Completed | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- I PNCA With Basal: Parent and Nurse Controlled Analgesics with basal
  Pain and standard side effect management for PNCA with basal method.: Comparing pain management and parent and nurse satisfaction with medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
- II PNCA w/o Basal: Parent and Nurse Controlled Analgesics without basal
  Pain and standard side effect management with PNCA without basal: Comparing pain management and parent nurse satisfaction with pain mediation delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
- III PRN Intermittent: Intermittent opioid administered IV on an "as needed" basis
  Pain and standard side effect management with IV on an as needed basis method.: Comparing pain management and parent and nurse satisfaction with pain medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol.
- Total: Total of all reporting groups
Arm/Group | I PNCA With Basal | II PNCA w/o Basal | III PRN Intermittent | Total
Number analyzed (Participants) | 22 | 30 | 28 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 30 | 28 | 80
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.5 [7.75 to 15.50] | 12 [9.75 to 15] | 12 [9 to 15] | 12 [9 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 11 | 34
  Male | 14 | 15 | 17 | 46
Region of Enrollment [Number; unit: participants]
  United States | 22 | 30 | 28 | 80

OUTCOME MEASURES:

1. Primary Outcome: Median Pain Score During Shift 1, as Measured With the Face, Legs, Activity, Cry, Consolability Scale
Description: Pain is measured with the Face, Legs, Activity, Cry, Consolability scale (FLACC) is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The median pain score over the first shift (24 hours) is reported.
Time Frame: First 24 hours on study
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- PNCA Without Basal: Parent and Nurse Controlled Analgesics without basal
  Pain and standard side effect management with PNCA without basal: Comparing pain management and parent nurse satisfaction with pain mediation delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol. PCA teaching will be done per Policy and Procedure.
- Intermittent Opioid on as Needed Basis: Intermittent opioid administered IV on an "as needed" basis
  Pain and standard side effect management with IV on an as needed basis method.: Comparing pain management and parent and nurse satisfaction with pain medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol.
Arm/Group | PNCA With Basal | PNCA Without Basal | Intermittent Opioid on as Needed Basis
Number analyzed (Participants) | 22 | 30 | 28
units on a scale | 1.0 [0.4 to 1.7] | 1.8 [0.2 to 3.0] | 1.5 [0.5 to 2.3]

2. Secondary Outcome: Number of Patients Requiring Naloxone for Respiratory Depression
Description: Number of patients requiring naloxone for respiratory depression (our most important side effect)
Time Frame: Daily, for up to 3 days
Measure: Count of Participants; unit: Participants
Groups:
- PRN Intermittent Opioids: Intermittent opioid administered IV on an "as needed" basis
  Pain and standard side effect management with IV on an as needed basis method.: Comparing pain management and parent and nurse satisfaction with pain medication delivery. Standard side effects of nausea, vomiting and pruritis can be expected although not always present. Protocol is in place to treat and manage these side effects.
  Only PAIN TEAM will be writing analgesic orders and will make medication adjustment per protocol.
Arm/Group | PNCA With Basal | PNCA Without Basal | PRN Intermittent Opioids
Number analyzed (Participants) | 22 | 30 | 28
Participants | 1 | 0 | 0

3. Secondary Outcome: Parent Satisfaction With the Administration Technique
Description: Parents were asked "Overall, how satisfied were you with the pain relief your child received after surgery?" Response options were: 1. Very Dissatisfied, 2. Dissatisfied, 3. Satisfied, 4. Very Satisfied. Responses were scored on a 1-4 scale, with Very Dissatisfied = 1; Dissatisfied = 2; Satisfied = 3; Very Satisfied = 4.
Time Frame: parents, once at the end of study
Population: Data was obtained from parents who completed the satisfaction survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I PNCA With Basal | II PNCA w/o Basal | III PRN Intermittent
Number analyzed (Participants) | 21 | 28 | 26
units on a scale | 1.32 (0.48) | 1.48 (0.57) | 1.65 (0.69)

ADVERSE EVENTS:
Arm/Group | I PNCA With Basal | II PNCA w/o Basal | III PRN Intermittent
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/27 | 0/34 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I PNCA With Basal (N=27) | II PNCA w/o Basal (N=34) | III PRN Intermittent (N=33)
respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pt's POX and respiratory rate decreased d/t parent not following protocol instructions. Naloxone administered, No negative sequele

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No